CLINICAL TRIAL: NCT05425004
Title: A Phase II Study of Cabozantinib for Patients With Recurrent or Progressive Meningioma
Brief Title: Cabozantinib for Patients With Recurrent or Progressive Meningioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KOT-002
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Meningioma
Keywords: Meningioma; central nervous system tumors; Recurrent meningioma; Progression meningioma
MeSH Terms: conditions — Meningioma; Central Nervous System Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Participants will self-administer cabozantinib 60 mg at the same time daily by mouth on a continuous 28-day schedule. Participants will continue to take this medication as long as they are deriving benefit from it without significant treatment-related toxicities.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib tablets are supplied as film coated tablets containing cabozantinib malate equivalent to 20 mg and 60 mg of cabozantinib and contain microcrystalline cellulose, lactose anhydrous, hydroxypropyl cellulose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate and Opadry® yellow. The 60 mg tablets are oval and the 20 mg tablets are round. Doses of 40 mg will comprise two 20-mg tablets.
  Other Names: XL184; Cometriq; Cabometyx; BMS907351

SUMMARY:
A Phase II Study of Cabozantinib for Patients with Recurrent or Progressive Meningioma

ELIGIBILITY:
Inclusion Criteria

1. Histologic (preferred) or radiologic diagnosis of meningioma. All World Health Organization (WHO) grades (I, II and III) are allowed.
2. All patients must have developed recurrent disease or progressive disease after receiving standard therapy (e.g., radiation or surgery) > 6 months ago or have been deemed ineligible to receive these therapies.
3. Karnofsky Performance Status ≥ 50.
4. Adequate hematologic function:

   1. Absolute Neutrophil Count ≥ 1.5 x 10^9 / L without granulocyte colony-stimulating factor support.
   2. Platelet Count ≥ 100 x 10^9 / L without transfusion.
   3. Hemoglobin ≥ 9 g/dL without transfusion within 7 days prior to screening assessment.
5. Adequate renal function: ≥ 30 ml/min according to the Cockcroft-Gault formula.
6. Adequate hepatic function including:

   1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN).
   2. Aspartate transaminase (AST) ≤ 3 x ULN without liver metastasis.
   3. Alanine transaminase (ALT) ≤ 3 x ULN without liver metastasis.
   4. AST or ALT ≤ 5 x ULN for patients with liver metastasis.
   5. Patients with known Gilbert's syndrome may be included if total bilirubin ≤ x 3 ULN.
7. Patients must have measurable disease by iRANO criteria
8. Women of childbearing potential must have negative serum pregnancy testing at screening. All women will be considered childbearing potential unless meeting criteria including:

   1. Achieved post-menopausal status as defined by cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and have follicular stimulation hormone showing postmenopausal state. Women who have been amenorrhoeic for ≥12 months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anorexia, low body weight, ovarian suppression, anti-estrogen therapy or other medically inducible reasons.
   2. Documented hysterectomy or bilateral oophorectomy surgery.
   3. Medically confirmed ovarian failure.
   4. Sexually active participants and their partners must agree to use medically. accepted methods of contraception during the study and for 4 months after discontinuing study treatment
9. Recovery of baseline CTCAE v5.0 Grade ≤1 toxicity related to prior study treatments unless adverse events are clinically non-significant per investigator's discretion and/or stable on supportive therapy if needed.
10. Patients must be willing and able to comply with trial protocol. This includes adhering to the treatment plan, scheduled visits, laboratory and other study procedures.
11. Serum albumin ≥ 2.8 g/dL.
12. Prothrombin time (PT)/International Normalized Ratio (INR) or partial thromboplastin time (PTT) test < 1.3x the laboratory ULN.

Exclusion Criteria

1. Prior treatment with cabozantinib.
2. Patients < 18 years old.
3. Patients who are pregnant or breast-feeding.
4. Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to the first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
5. Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
6. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) with 2 weeks before first dose of study treatment.
7. Ejection fraction (EF) ≤ 50% by echocardiogram (ECHO). Multi-gated acquisition scan (MUGA) should be obtained to estimate EF if quality of ECHO is insufficient.
8. Prior history of hypertensive encephalopathy at any time.
9. History of congenital QT syndrome.
10. Correct QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 14 days of study registration. If initial QTcF is >500 ms, two additional EKGs separated by at least 3 minutes should be performed, and if average of these consecutive results is QTcF is ≤ 500 ms, patient is eligible.
11. Unstable cardiac arrhythmia within 6 months prior to study registration date.
12. Urine Protein-to-Creatinine ratio (UPCR) >1 mg/mg or 24-hour urine protein > 1 gram.
13. History of bleeding diathesis or significant unexplained coagulopathy (e.g., in the absence of anticoagulation).
14. Clinical signs or symptoms of gastrointestinal obstruction requiring parenteral hydration, nutrition or feeding tube.
15. Uncontrolled effusion management (pleural effusion, pericardial effusion or ascites) requiring recurrent drainage procedures.
16. Active infection requiring parenteral antibiotic therapy.
17. History of either positive hepatitis C virus (HCV) RNA viral load or detectable anti-HCV antibody; hepatitis B virus (HBV) infection with HBV surface antigen detection and/or positive HBV DNA viral load.
18. Serious non-healing wound, ulcer, or bone fracture requiring intervention within 28 days prior to study registration date.
19. Known hypersensitivity to cabozantinib or any component in formulation.
20. Inability to swallow capsules, known intolerance to cabozantinib or its excipients, known malabsorption syndrome, or other conditions which impair intestinal absorption.
21. Other severe acute or chronic medical conditions, which may increase study risk per treating investigator's discretion.
22. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

    1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
23. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    1. Cardiovascular disorders:
    2. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    3. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    4. Stroke [including transient ischemic attack (TIA)], myocardial infarction (MI), or other ischemic event, or thromboembolic event [e.g., deep venous thrombosis (DVT), pulmonary embolism (PE)] within 6 months before first dose of study treatment.
    5. Subjects with a diagnosis of incidental, sub-segmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment.
    6. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:
    7. The subject has evidence of any concurrent malignancy invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    8. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
24. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
25. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease from another malignancy.
26. Other clinically significant disorders that would preclude safe study participation.

    1. Serious non-healing wound/ulcer/bone fracture.
    2. Uncompensated/symptomatic hypothyroidism.
    3. Moderate to severe hepatic impairment (Child-Pugh B or C).
27. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 months
  Proportion of participants who from start of treatment to 6-months are free from objective tumor progression or death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Proportion of participants with confirmed complete response (CR) or partial response (PR) assessed by Immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria, relative to the total population of patients enrolled who initiate therapy.
Overall survival (OS) | 2 years
  Overall Survival (OS): duration of time from start of treatment until death from any cause. Patients lost-to follow up will be censored at last valid assessment.
Proportion of participants with adverse events | 2 years
  Proportion of participants who develop adverse events assessed by CTCAE v5.0 criteria.
Quality of life (QOL) | 2 years
  QOL will be measured by Functional Assessment of Cancer Therapy-Brain (FACT-Br) Version 4. The FACT-Br questionnaire is a 23-item survey, participants then rate each item on a Likert scale from 0 "not at all" to 4 "very much", and overall, higher ratings are suggestive of better quality of life.
  QOL will be assessed at the baseline, day 1 of every cycle (treatment days, every 4 weeks on 28-day cycle, and every 6 weeks on 42-day cycle).

CONTACTS AND LOCATIONS:
Overall Officials: Yazmin Odia, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (3):
- United States (3):
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rogers CL, Won M, Vogelbaum MA, Perry A, Ashby LS, Modi JM, Alleman AM, Galvin J, Fogh SE, Youssef E, Deb N, Kwok Y, Robinson CG, Shu HK, Fisher BJ, Panet-Raymond V, McMillan WG, de Groot JF, Zhang P, Mehta MP. High-risk Meningioma: Initial Outcomes From NRG Oncology/RTOG 0539. Int J Radiat Oncol Biol Phys. 2020 Mar 15;106(4):790-799. doi: 10.1016/j.ijrobp.2019.11.028. Epub 2019 Nov 29. PMID 31786276
- [Background] Jaaskelainen J, Haltia M, Servo A. Atypical and anaplastic meningiomas: radiology, surgery, radiotherapy, and outcome. Surg Neurol. 1986 Mar;25(3):233-42. doi: 10.1016/0090-3019(86)90233-8. PMID 3945904
- [Background] Perry A, Scheithauer BW, Stafford SL, Lohse CM, Wollan PC. "Malignancy" in meningiomas: a clinicopathologic study of 116 patients, with grading implications. Cancer. 1999 May 1;85(9):2046-56. doi: 10.1002/(sici)1097-0142(19990501)85:93.0.co;2-m. PMID 10223247
- [Background] Perry A, Stafford SL, Scheithauer BW, Suman VJ, Lohse CM. Meningioma grading: an analysis of histologic parameters. Am J Surg Pathol. 1997 Dec;21(12):1455-65. doi: 10.1097/00000478-199712000-00008. PMID 9414189
- [Background] Preusser M, Brastianos PK, Mawrin C. Advances in meningioma genetics: novel therapeutic opportunities. Nat Rev Neurol. 2018 Feb;14(2):106-115. doi: 10.1038/nrneurol.2017.168. Epub 2018 Jan 5. PMID 29302064
- [Background] Yun S, Koh JM, Lee KS, Seo AN, Nam KH, Choe G. Expression of c-MET in Invasive Meningioma. J Pathol Transl Med. 2015 Jan;49(1):44-51. doi: 10.4132/jptm.2014.10.13. Epub 2015 Jan 15. PMID 25812657
- [Background] Kaley TJ, Wen P, Schiff D, Ligon K, Haidar S, Karimi S, Lassman AB, Nolan CP, DeAngelis LM, Gavrilovic I, Norden A, Drappatz J, Lee EQ, Purow B, Plotkin SR, Batchelor T, Abrey LE, Omuro A. Phase II trial of sunitinib for recurrent and progressive atypical and anaplastic meningioma. Neuro Oncol. 2015 Jan;17(1):116-21. doi: 10.1093/neuonc/nou148. Epub 2014 Aug 6. PMID 25100872
- [Background] Chevreau C, Ravaud A, Escudier B, Amela E, Delva R, Rolland F, Tosi D, Oudard S, Blanc E, Ferlay C, Negrier S; French Group on Renal Cancer. A phase II trial of sunitinib in patients with renal cell cancer and untreated brain metastases. Clin Genitourin Cancer. 2014 Feb;12(1):50-4. doi: 10.1016/j.clgc.2013.09.008. Epub 2013 Sep 28. PMID 24268852
- [Background] Ma PC, Tretiakova MS, MacKinnon AC, Ramnath N, Johnson C, Dietrich S, Seiwert T, Christensen JG, Jagadeeswaran R, Krausz T, Vokes EE, Husain AN, Salgia R. Expression and mutational analysis of MET in human solid cancers. Genes Chromosomes Cancer. 2008 Dec;47(12):1025-37. doi: 10.1002/gcc.20604. PMID 18709663
- [Background] Wen PY, Drappatz J, de Groot J, Prados MD, Reardon DA, Schiff D, Chamberlain M, Mikkelsen T, Desjardins A, Holland J, Ping J, Weitzman R, Cloughesy TF. Phase II study of cabozantinib in patients with progressive glioblastoma: subset analysis of patients naive to antiangiogenic therapy. Neuro Oncol. 2018 Jan 22;20(2):249-258. doi: 10.1093/neuonc/nox154. PMID 29016998
- [Background] Choueiri TK, Escudier B, Powles T, Mainwaring PN, Rini BI, Donskov F, Hammers H, Hutson TE, Lee JL, Peltola K, Roth BJ, Bjarnason GA, Geczi L, Keam B, Maroto P, Heng DY, Schmidinger M, Kantoff PW, Borgman-Hagey A, Hessel C, Scheffold C, Schwab GM, Tannir NM, Motzer RJ; METEOR Investigators. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1814-23. doi: 10.1056/NEJMoa1510016. Epub 2015 Sep 25. PMID 26406150
- [Background] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Background] Escudier B, Powles T, Motzer RJ, Olencki T, Aren Frontera O, Oudard S, Rolland F, Tomczak P, Castellano D, Appleman LJ, Drabkin H, Vaena D, Milwee S, Youkstetter J, Lougheed JC, Bracarda S, Choueiri TK. Cabozantinib, a New Standard of Care for Patients With Advanced Renal Cell Carcinoma and Bone Metastases? Subgroup Analysis of the METEOR Trial. J Clin Oncol. 2018 Mar 10;36(8):765-772. doi: 10.1200/JCO.2017.74.7352. Epub 2018 Jan 8. PMID 29309249
- [Background] Choueiri TK, Hessel C, Halabi S, Sanford B, Michaelson MD, Hahn O, Walsh M, Olencki T, Picus J, Small EJ, Dakhil S, Feldman DR, Mangeshkar M, Scheffold C, George D, Morris MJ. Cabozantinib versus sunitinib as initial therapy for metastatic renal cell carcinoma of intermediate or poor risk (Alliance A031203 CABOSUN randomised trial): Progression-free survival by independent review and overall survival update. Eur J Cancer. 2018 May;94:115-125. doi: 10.1016/j.ejca.2018.02.012. Epub 2018 Mar 20. PMID 29550566
- [Background] Abou-Alfa GK, Meyer T, Cheng AL, El-Khoueiry AB, Rimassa L, Ryoo BY, Cicin I, Merle P, Chen Y, Park JW, Blanc JF, Bolondi L, Klumpen HJ, Chan SL, Zagonel V, Pressiani T, Ryu MH, Venook AP, Hessel C, Borgman-Hagey AE, Schwab G, Kelley RK. Cabozantinib in Patients with Advanced and Progressing Hepatocellular Carcinoma. N Engl J Med. 2018 Jul 5;379(1):54-63. doi: 10.1056/NEJMoa1717002. PMID 29972759
- [Background] Foxx-Lupo WT, Sing S, Alwan L, Tykodi SS. A Drug Interaction Between Cabozantinib and Warfarin in a Patient With Renal Cell Carcinoma. Clin Genitourin Cancer. 2016 Feb;14(1):e119-21. doi: 10.1016/j.clgc.2015.09.015. Epub 2015 Oct 3. No abstract available. PMID 26549824
- [Background] Raizer JJ, Fitzner KA, Jacobs DI, Bennett CL, Liebling DB, Luu TH, Trifilio SM, Grimm SA, Fisher MJ, Haleem MS, Ray PS, McKoy JM, DeBoer R, Tulas KM, Deeb M, McKoy JM. Economics of Malignant Gliomas: A Critical Review. J Oncol Pract. 2015 Jan;11(1):e59-65. doi: 10.1200/JOP.2012.000560. Epub 2014 Dec 2. PMID 25466707
- [Background] Grimm SA, Chamberlain MC. Bevacizumab and other novel therapies for recurrent oligodendroglial tumors. CNS Oncol. 2015;4(5):333-9. doi: 10.2217/cns.15.27. Epub 2015 Oct 28. PMID 26509217
- [Background] Shih KC, Chowdhary S, Rosenblatt P, Weir AB 3rd, Shepard GC, Williams JT, Shastry M, Burris HA 3rd, Hainsworth JD. A phase II trial of bevacizumab and everolimus as treatment for patients with refractory, progressive intracranial meningioma. J Neurooncol. 2016 Sep;129(2):281-8. doi: 10.1007/s11060-016-2172-3. Epub 2016 Jun 16. PMID 27311730
- See also: Miami Cancer Institute — https://cancer.baptisthealth.net/